CLINICAL TRIAL: NCT01299233
Title: Reproducibility of RNFL Circle Scans With ART-Function of Heidelberg Spectralis SD-OCT Software Version 5.3
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: ART-OCT
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-12

CONDITIONS: Glaucoma Patients and Healthy Controls
MeSH Terms: interventions — Proton Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control group: age matched healthy controls
  Interventions: Device: Spectralis® SD-OCT, Heidelberg Engineering GmbH, H
- Glaucoma: patients with diagnosis of primary open angle glaucoma
  Interventions: Device: Spectralis® SD-OCT, Heidelberg Engineering GmbH, H

INTERVENTIONS:
Device: Spectralis® SD-OCT, Heidelberg Engineering GmbH, H — Measurement of the peripapillar nerve fiber layer with different settings of ART

SUMMARY:
To assess the improvement in reproducibility of 100 vs. 16 averaged images by Automatic Real Time (ART) using Spectralis™ Spectral Domain-Optical Coherence Tomography (SD-OCT, Heidelberg Engineering GmbH, Heidelberg, Germany) in retinal nerve fiber layer thickness (RNFL) circle scan-measurements.

* Trial with medical device

ELIGIBILITY:
Inclusion criteria:

for both groups (glaucoma study group and control group): men and women of at least 50 years of age

for the glaucoma study group: diagnosis of primary open angle glaucoma (POAG)

Exclusion criteria:

for both groups (glaucoma study group and control group):

* less then 18 years of age
* any pathology of the central retina
* any optic nerve disorder other then glaucoma
* retinal vascular disorder

for the glaucoma study group: other glaucoma diagnosis then primary open angle glaucoma

for the control group: any diagnosis of glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients and controls are selected out of our primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
COV | T0

CONTACTS AND LOCATIONS:
Overall Officials: Jens Funk, Prof. MD, Principal Investigator — University Hospital Zurich, Ophtalmic Clinic
Locations (1):
- University Hospital Zurich, Ophthalmic Clinic, Zurich, Canton of Zurich, Switzerland